CLINICAL TRIAL: NCT04859738
Title: The Effect of Topical Lidocaine and Benzocaine on Pain and Injection Satisfaction in Peripheral Intravenous Catheter Applications
Brief Title: The Effect of Lidocaine and Benzocaine on Pain and Injection Satisfaction in Peripheral Intravenous Catheter Application
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ali Kaplan, Lecturer, TC Erciyes University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Ali KAPLAN Erciyes University
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Peripheral Intravenous Catheterization Application
Keywords: Peripheral intravenous catheterization; pain; injection satisfaction; pharmacological method; lidocaine; benzocaine
MeSH Terms: conditions — Pain | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: During the data collection, 120 individuals who met the inclusion criteria and were selected with the randomization list created on the computer constituted the sample of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experiment I Group (Lidocaine Spray) (Experimental): Lidocaine Spray was applied to Experiment I group before peripheral intravenous catheter application.
  Interventions: Drug: Lidocaine Spray
- Experiment II Group (Benzokain Sprey) (Experimental): Benzokain Sprey was applied to Experiment II group before peripheral intravenous catheter application.
  Interventions: Drug: Benzokain Sprey
- Placebo Group (Placebo Comparator): Alcohol was administered to the placebo group prior to peripheral intravenous catheter application.
  Interventions: Other: Alcohol

INTERVENTIONS:
Drug: Lidocaine Spray — Individuals who met the research criteria and signed the informed consent form were numbered according to the order in which they came to the hospital. Later, the numbered individuals were assigned to the study groups according to the randomization list created in the computer environment.
  Lidocaine Spray was applied 60 seconds before to the area where the peripheral intravenous catheter application of the patients in the Experiment I Group (Lidocaine Spray) will be performed. After waiting 60 seconds, peripheral intravenous catheter application was performed.
  The nurse responsible for data collection measured blood pressure, pulse rate and peripheral oxygen saturation values 5 minutes before and just after the application with a finger-type pulse oximeter.
  After performing peripheral intravenous catheterization, the pain level felt by the individual during the procedure and the injection satisfaction level values were taken and recorded on the Case Report Form by the nurse.
  Arms: Experiment I Group (Lidocaine Spray)
Drug: Benzokain Sprey — Individuals who met the research criteria and signed the informed consent form were numbered according to the order in which they came to the hospital. Later, the numbered individuals were assigned to the study groups according to the randomization list created in the computer environment.
  Benzocaine Spray was applied 60 seconds before to the area where the peripheral intravenous catheter will be applied to the patients in the Experiment II Group (Benzocaine Spray). After waiting 60 seconds, peripheral intravenous catheter application was performed.
  The nurse responsible for data collection measured blood pressure, pulse rate and peripheral oxygen saturation values 5 minutes before and just after the application with a finger-type pulse oximeter.
  After performing peripheral intravenous catheterization, the pain level felt by the individual during the procedure and the injection satisfaction level values were taken and recorded on the Case Report Form by the nurse.
  Arms: Experiment II Group (Benzokain Sprey)
Other: Alcohol — Individuals who met the research criteria and signed the informed consent form were numbered according to the order in which they came to the hospital. Later, the numbered individuals were assigned to the study groups according to the randomization list created in the computer environment.
  In patients in the placebo group, alcohol was sprayed 60 seconds before the area where the peripheral intravenous catheter will be applied. After waiting 60 seconds, peripheral intravenous catheter application was performed.
  The nurse responsible for data collection measured blood pressure, pulse rate and peripheral oxygen saturation values 5 minutes before and just after the application with a finger-type pulse oximeter.
  After performing peripheral intravenous catheterization, the pain level felt by the individual during the procedure and the injection satisfaction level values were taken and recorded on the Case Report Form by the nurse.
  Arms: Placebo Group

SUMMARY:
Objective: This research was conducted as a randomized controlled, double-blind experimental study to determine the effect of topical lidocaine and benzocaine on patient's pain and injection satisfaction before peripheral intravenous catheter application.

Study Design: The study was completed with 120 individuals who were treated in the green area of a University Hospital Emergency Service and met the inclusion criteria of the study. In collecting research data; Case Report Form (ORF), Baseline Algometer (66 Lb / 30 Kg) and Informed Consent Form were used. Lidocaine Spray, Benzocaine Spray and Alcohol were used in research groups.

DETAILED DESCRIPTION:
Objective: This research was conducted as a randomized controlled, double-blind experimental study to determine the effect of topical lidocaine and benzocaine on patient's pain and injection satisfaction before peripheral intravenous catheter application.

Study Design: The study was completed with 120 individuals who were treated in the green area of a University Hospital Emergency Service and met the inclusion criteria of the study. Ethics committee approval, Turkey Pharmaceuticals and Medical Devices Agency clinical research permission, institutional permission and written informed consent from individuals were obtained in the study. In collecting research data; Case Report Form (ORF), Baseline Algometer (66 Lb / 30 Kg) and Informed Consent Form were used. Lidocaine Spray, Benzocaine Spray and Alcohol were used in research groups. Private health insurance was provided for all patients included in the study for complications arising from the procedure. The data obtained from the research were evaluated in computer environment using IBM SPSS Statistics 23.0 statistics package program.

ELIGIBILITY:
Inclusion Criteria:

* Can speak and understand Turkish,
* Over the age of 18,
* Under the age of 65,
* Located in the green area of Erciyes University Emergency Service,
* Having orientation in place and time,
* Not using psychiatric medication due to any psychiatric illness,
* Not using central nervous system drugs,
* Does not have any known chronic disease,
* No vision or hearing problems,
* No signs of phlebitis, scar tissue, dermatitis, incision or infection in the area to be operated,
* Does not have pain anywhere on the body that will affect the result of the study and whose visual comparison scale pain score is zero at the time of application
* No experience of IV catheter application in the last month,
* Not taking analgesic in the last 24 hours,
* Intravenous drug treatment is ordered,
* With Baseline Algometer device, the average pressure pain threshold is 8-16 pounds (Lb),
* Individuals who volunteered to participate in the study and signed the written consent form were included in the study.

Exclusion Criteria:

* Not wanting to participate in the study,
* A history of sensitivity to the study drug or related drugs or any drug excipient,
* Having clinically significant vital signs,
* Stating that he / she is addicted to alcohol and drugs,
* Those who were incompetent or unwilling to comply with the study protocol or who stated that they experienced difficulties in the procedures related to the study (eg establishing vascular access before) were not included in the study.
* In patients who developed IV catheter complications (swelling of the vascular access, hematoma) during the study,
* In patients whose IV catheter insertion cannot be performed at the first time,
* The study was terminated in patients who wanted to leave the study anywhere in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Pain level (Visual Analog Scale) | Evaluation was made immediately after application.
  Visual Analog Scale is a scale used to measure the severity of pain. It is used to numerically convert the pain value that cannot be measured numerically. The two end definitions of the pain parameter are written on both ends of a 100 mm line and the patient is asked to indicate where his condition is appropriate by drawing a line, placing a dot or marking on this line. It is a 100 mm (10 cm) ruler that can be used horizontally and vertically, with painlessness on one end and the most severe pain on the other. "0 mm" means painlessness, "100 mm" means the most severe pain. The individual indicates the severity of the pain he feels on this scale. In line with these data, horizontally prepared Visual Analog Scale was used in this study to determine the severity of pain felt by patients during peripheral IV catheter injection. Pain severity score measurements were evaluated in mm.

SECONDARY OUTCOMES:
Injection Satisfaction Scale | Evaluation was made immediately after application.
  It is a scale created to determine the satisfaction status of patients due to injection after peripheral IV catheter injection. The two tip definitions of the injection satisfaction parameter are written on both ends of a 100 mm line and the patient is asked to indicate where his condition is appropriate by drawing a line, point or mark on this line. It is a 100 mm (10 cm) ruler that can be used horizontally and vertically, with one end saying "I'm not satisfied at all, but very satisfied" on the other. "0mm" means not satisfied at all, "100mm" means very satisfied. The individual determines the degree of satisfaction with the injection felt on this scale. In line with the above findings, horizontally prepared Injection Satisfaction Scale was used in this study to determine the injection satisfaction levels of patients due to peripheral intravenous catheter injection application. Injection satisfaction levels score measurements were evaluated in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No